CLINICAL TRIAL: NCT05775601
Title: A Phase 1, Open-label Study to Evaluate the Biodistribution and Safety of 18F-LY3950321 (18F-MNI-1256) in Healthy Subjects
Brief Title: 18F-LY3950321-01 Biodistribution and Safety Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-LY3950321-01
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Diagnostic Agent Adverse Reaction; Radiation Exposure
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-LY3950321 Whole Body Dosimetry (Experimental)
  Interventions: Drug: 18F-LY3950321; Procedure: PET Scan

INTERVENTIONS:
Drug: 18F-LY3950321 — 3 millicuries (±1 mCi)
  Other Names: 18F-MNI-1256
Procedure: PET Scan — positron emission tomography (PET) scan

SUMMARY:
18F-LY3950321 (also known as 18F-MNI-1256) is a radiolabeled positron emission tomography (PET) tracer targeting granzyme B. The overall goal of this protocol is to evaluate the safety, tolerability, and radiation dosimetry of 18F-LY3950321.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no clinically relevant finding on physical examination at Screening and upon reporting to the clinic for the Imaging Visit.
* Female subjects must not be of childbearing potential, or if they are of childbearing potential to agree to use contraception and not donate eggs.
* Male subjects with their partners of childbearing potential must commit to the use of 2 methods of contraception, 1 of which is a barrier method for male subjects for the study duration and 90 days after study completion.
* Male subjects must not donate sperm for the study duration and for 90 days after study completion.

Exclusion Criteria:

* Current or prior history of any alcohol or drug abuse in the past 2 years.
* Currently exposed to nicotine products or had regular nicotine exposure within a six-month period, to be verified by urine cotinine screening.
* ECG or Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Known history of hypersensitivity, including hypersensitivity to the active substances used for 18F-LY3950321 or derivatives, or to any of the associated excipients.
* Subject has received an investigational drug within 30 days or five half-lives prior to Day 1, whichever is longer.
* Prior participation in other research protocols or clinical care during the past year that would result in radiation exposure to an effective radiation dose exceeding the acceptable annual limit established by the US Federal Guidelines (effective dose of 50 milliSieverts, including the procedures in this clinical protocol).
* Pregnant, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* Use of any prescription drugs (except approved forms of birth control) or herbal supplements, within 4 weeks prior to Day 1.
* Use of any over-the-counter (OTC) medication or dietary supplements (vitamins included) within 2 weeks prior to Day 1.
* Subject is, in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
18F-LY3950321 Whole Body Effective Dose | injection to 4 hours postdose
  Radiation dose estimates. Distribution data will be utilized in the MIRD calculations of target organ radiation absorbed dose with correction from urine assays and standard GI kinetic models in Organ Level Internal Dose Assessment (OLINDA). Standard Medical Internal Radiation Dose (MIRD) assumptions will be incorporated in dosimetry models for determination of radiation absorbed doses in target organs and whole-body.

CONTACTS AND LOCATIONS:
Overall Officials: Avid Medical Director, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (1):
- Invicro, LLC, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stabin MG, Sparks RB, Crowe E. OLINDA/EXM: the second-generation personal computer software for internal dose assessment in nuclear medicine. J Nucl Med. 2005 Jun;46(6):1023-7. PMID 15937315
- [Background] International Commission on Radiological Protection. Human alimentary tract model for radiological protection. ICRP Publication 100. A report of The International Commission on Radiological Protection. Ann ICRP. 2006;36(1-2):25-327, iii. doi: 10.1016/j.icrp.2006.03.004. PMID 17188183
- [Background] Harrison J, Lopez PO. Use of effective dose in medicine. Ann ICRP. 2015 Jun;44(1 Suppl):221-8. doi: 10.1177/0146645315576096. Epub 2015 Mar 25. PMID 25816282